CLINICAL TRIAL: NCT00399178
Title: A Randomised Open Controlled Parallel Group Multicenter Study to Evaluate the Efficacy and Safety of Norspan Versus Tiparol Retard in Subjects With Chronic Moderate to Severe OA Pain of the Hip and/or Knee.
Brief Title: A Randomised Open Controlled Parallel Group Study Comparing Norspan and Tramadol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma AB (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-003233-32; BUP4009
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2007-08-17 (Estimated); Status verified 2006-11

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Norspan versus Tramadol; Randomised; Efficacy and safety; OA pain of the hip and/or knee
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Drug: Transdermal delivery system

SUMMARY:
To evaluate the efficacy and safety of Norspan versus Tiperol Retard among OA patients who are sub-optimally treated with current analgesic. Those patients may benefit from treatment with a long lasting analgesic.

ELIGIBILITY:
Inclusion Criteria:

* OA diagnosis
* BS11 greater than or equal to 4 at base line
* Not adequately pain relieved with 4,000 mg paracetamol daily

Exclusion Criteria:

* Treated with high potent opioids for their OA pain
* Treated with a regular dose for greater than one week of Tramadol, Codeine or dextropropoxifene during the last three months
* Other chronic conditions requiring frequent analgesic therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2006-11; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Box Scale 11 pain scores for pain on average during the last week then mean change from base line to completion. BS11 is recorded daily by the patients in a diary.

SECONDARY OUTCOMES:
Rescue medication recorded daily by patients. Sleep disturbance and quality of sleep. Patients global assessment of pain relief, investigators global assessment of pain relief, patients preference, WOMAC OA index, EuroQoL EQ-5D.

CONTACTS AND LOCATIONS:
Overall Officials: M Karlsson, Med, Principal Investigator
Locations (1):
- Dr Mats Karlsson, Falköping, Parkgatan 6C, Sweden